CLINICAL TRIAL: NCT03376035
Title: Pilot Study Assessing Cutaneous Breast Temperature in the Setting of Mastectomy and Reconstruction
Brief Title: Pilot Study Assessing Breast Temperature in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00084743
Record Dates: First submitted 2017-12-05; First posted 2017-12-18 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Breast Reconstruction

STUDY DESIGN:
Intervention Model Description: Determine skin temperature after breast reconstruction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Unilateral breast reconstruction (Active Comparator): Temperature measurements are obtained from the reconstructed breast and compared to the non-reconstructed breast.
  Interventions: Other: Temperature measurement of breast
- Bilateral breast reconstruction (Experimental): Temperature measurements are obtained from both reconstructed breasts and the core temperature is measured as well for comparison.
  Interventions: Other: Temperature measurement of breast

INTERVENTIONS:
Other: Temperature measurement of breast — Multiple measurements will be obtained from the ear, chest, breast, abdomen, and hands.

SUMMARY:
Our investigators plan to measure the skin on the breast six months after breast reconstruction. The non-reconstructed breast will be used as the control for subject with unilateral reconstruction only. For those who have BILATERAL reconstruction, a core temperature will be obtained from the ear.

DETAILED DESCRIPTION:
Many factors influence outcomes following mastectomy and breast reconstruction. Cutaneous sensation, degree of scar formation, nipple projection and overall appearance are well correlated with patient satisfaction. However, very little data exists on the importance of skin temperature after mastectomy and reconstruction. Our investigators have noted that a number of patients report their reconstructed breast is cold and relate this as a source of dis-satisfaction. In these patients, it is unclear if 1) the reconstructed breast skin is cold and if so 2) can something can be done to improve this. Our investigators hypothesize that cutaneous breast temperature may be altered after mastectomy and reconstruction. This may be dependent on the reconstruction technique and other patient factors. In this pilot study, our investigators aim to establish techniques for evaluating cutaneous breast temperature following mastectomy and reconstruction. Our investigators hope to establish baseline data to develop an understanding of breast skin temperature after mastectomy and reconstruction.

Our long-term goals are to evaluate how cutaneous breast temperature may contribute to patient satisfaction. Our investigators also hope to determine which patients are at risk for developing a cold breast after surgery. Finally, our investigators will setup a prospective trial evaluating techniques to correct this problem and improve patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* For post-reconstruction patients: all patients who have undergone mastectomy and breast reconstruction at Duke and are seen in clinic no sooner than 3 months after reconstruction and no more than 5 years after reconstruction.

Exclusion Criteria:

* Metastatic malignancy of any kind.
* Subjects with a history of breast implant augmentation prior to mastectomy and reconstruction.
* Subjects who cannot give an informed consent.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 52 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
Change in skin temperature after breast reconstruction | 6 months after surgery
  Temperature measurements

CONTACTS AND LOCATIONS:
Overall Officials: Scott Hollenbeck, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No